CLINICAL TRIAL: NCT00747942
Title: Intervention Program for Physically Inactive and Overweight Immigrant Women From the Middle East and Latin America Living in Sweden
Brief Title: Support for Increased Physical Activity (Stöd Till Aktivare Motion)
Acronym: STAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Kristina Sundqvist, Professor, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-1165
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Overweight
Keywords: overweight; physical inactivity; physical fitness; lifestyle change
MeSH Terms: conditions — Overweight; Sedentary Behavior | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): exercise referral to lifestyle activities at the level of moderate intensity without support
- B (Active Comparator): Exercise referral combined with individual support, access to structured group exercise programs, and motivational support
  Interventions: Behavioral: Support for Increased Physical Activity

INTERVENTIONS:
Behavioral: Support for Increased Physical Activity — Exercise referral combined with individual support, access to structured group exercise programs, and motivational support
  Other Names: STAM; Stöd Till Aktivare Motion
  Arms: B

SUMMARY:
The purpose of this study is to improve and analyze the level of physical activity in immigrant women from the Middle East and Latin America living in Sweden. The investigators will also investigate if glucose, insulin, and lipid metabolism; stress-related hormone production; and subclinical inflammatory activity are affected by the intervention. The follow-up period is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age 25 through 64 years
* Physical inactivity
* BMI > 25
* Immigrant to Sweden from either the Middle East or Latin America

Exclusion Criteria:

* Diabetes mellitus type I
* Ischemic heart disease
* Disability that interferes with the ability to participate in lifestyle-related physical activity

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The relative effectiveness of two physical activity programs in affecting glucose metabolism, lipid metabolism and stress-related hormone production | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundquist, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Center for Family and Community Medicine, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Derived] Sundquist J, Hagstromer M, Johansson SE, Sundquist K. Effect of a primary health-care-based controlled trial for cardiorespiratory fitness in refugee women. BMC Fam Pract. 2010 Aug 2;11:55. doi: 10.1186/1471-2296-11-55. PMID 20678219
- See also: Web page of sponsoring organization — http://www.cefam.se